CLINICAL TRIAL: NCT03298464
Title: A Phase 1B, Single Center, Randomized, Open Label, Parallel Group Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single NGM313 Dose or Daily Oral Pioglitazone in Obese Participants With Insulin Resistance and Increased Liver Fat
Brief Title: Study of NGM313 in Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0202
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Obese
MeSH Terms: conditions — Obesity | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NGM313 (Experimental)
  Interventions: Biological: NGM313
- Pioglitazone (Active Comparator)
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Biological: NGM313 — Subcutaneous injection
  Arms: NGM313
Drug: Pioglitazone — White to off-white round tablet
  Arms: Pioglitazone

SUMMARY:
The purpose of the study is to evaulate the safety, tolerability, and efficacy of NGM313 in obese participants

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 30-43 kg/m2
* Waist circumference > 40 inches in males or > 30 inches in females
* Normal ECG readings

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of any known Congestive heart failure (CHF)
* History of macrovascular disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of whole body insulin sensitivity measured as insulin sensitivity index (M and Si) following intravenous insulin administration | 28 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Prosciento, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No